CLINICAL TRIAL: NCT06375863
Title: QT Changes in Geriatric Patients: a Comparison of Spinal and General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sinan Uzman, associate prof, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 44-2023
Record Dates: First submitted 2024-03-22; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia, Spinal; Sevoflurane; Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal anesthesia (Other): patients who scheduled lower abdominal or urological surgery under spinal anesthesia older than 65 years
  Interventions: Diagnostic Test: QT and QTc interval
- general anesthesia (Other): patients who scheduled lower abdominal or urological surgery under general anesthesia older than 65 years
  Interventions: Diagnostic Test: QT and QTc interval

INTERVENTIONS:
Diagnostic Test: QT and QTc interval — measuring of QT and QTc on ECG

SUMMARY:
QT interval, defined as the time between the beginning of the QRS complex and the end of the T wave in electrocardiography (ECG), is an indicator of depolarization and repolarization of the myocardium.11 Prolongation of the heart rate corrected QT (QTc) interval reflects electrical instability of ventricles and is associated with life-threatening ventricular arrhythmias, including torsade de pointes, ventricular fibrillation and sudden cardiac death.

Spinal anesthesia can cause profound prolongation of the QTc interval due to disparity between lumbar and thoracic sympathetic activity following subarachnoid block. Meanwhile inhalational anesthetics, sevoflurane, isoflurane, and desflurane are known to prolong QTc interval and intravenous anesthetics such as propofol, thiopental, etomidate and ketamin can also cause remarkable prolongation of the QTc interval. Moreover laryngoscopy and intubation may contribute to prolongation of the QTc interval because of the sympathetic stimulation.

Over the years it has been occurred an increase in the proportion of elderly population requiring surgical anesthesia. The incidence of ventricular arrhythmias increases in advancing age even in the absence of underlying heart disease and elderly patients have reduced physiological functions and poor tolerance to anesthesia. However the choice of anesthesia type is critical in this population.

To the best of knowledge, there was no published study to compare spinal anesthesia and inhalational anesthesia in elderly patients with regard to the QT interval changes. Investigators aimed to investigate the effects of spinal anesthesia on QT, QTc intervals and to compare general anesthesia with sevofluran in elderly patients.

DETAILED DESCRIPTION:
Investigators designed a prospective, randomized trial to compare spinal and general anesthesia in elderly patients on the effects of QT interval changes. The study protocol was approved by the Health Science University Haseki Training and Research Hospital Ethics Committee, Istanbul, Turkey (date: 03/29/2023 and number: 44-2023). This study was conducted according to the Declaration of Helsinki, and written informed consent was obtained from all patients. The study was performed at a tertiary referral hospital with 700 beds in Istanbul, Turkey between 03/29/2023-05/29/2023.

The patients who will undergo lower abdominal or extremity surgery and urological surgery older than 65 years will be included in this study. The exclusion criteria are as follows: any preoperative ECG abnormalities, QTc interval > 440 ms, family history of long QT syndome, use of any medications known to affect the QTc interval, serum electrolyte abnormalities, any contraindications for spinal anesthesia (e.g. coagulation disorders), unstable angina pektoris, chronic obstructive pulmonary disease, hepatic or renal failure, American Society of Anesthesiologists (ASA) physical classification status > III, pregnancy and obesity (BMI > 30).

Participants will be divided into two groups: the spinal anesthesia (group S) and general anesthesia (group G). Randomization and group allocations will be performed by a researcher who did not participate the collection of data.

In the preoperative care unit all patients will receive 10 ml/kg Ringer's lactate solution via a peripheral vein over 30 minutes. In the operating room premedication will be obtained with 0.015 mg/kg of midazolam and 1 µg/kg fentanyl intravenously.

In group G, a 2.0 mg/kg propofol injection will be used for the induction of anesthesia and facilitating of endotracheal intubation was provided with 0.6 mg/kg rocuronium. After the intubation the patients will be ventilated with a 6-8 ml/kg of tidal volume in volume control ventilation (VCV) mode with an anesthesia machine (Dräger Primus, Dräger Medical Systems, Inc. Danvers, MA, USA). Frequency of respiration will be adjusted to maintain PET CO2 at 32-36 mm Hg. Maintenance of anesthesia will be provided with sevoflurane (1.5-2%) in an oxygen-air mixture (FiO2 = 0.4) and 0.015 mg/kg rocuronium as needed. At the end of the surgery residual neuromuscular block will be antagonized with 4 mg/kg sugammedex.

In group S, spinal anesthesia will be performed in the sitting position at the level of L3-4 or L4-5 using a 25-gauge Whitacre (pencil point) spinal needle after the obtaining strict sterile conditions and local anesthesia with intradermal lidocaine hydrochloride 1%. Hyperbaric bupivacaine (Marcaine Spinal 0.5% Heavy; AstraZeneca, Turkey) 3-4 mL of 0.5% will be injected to the subarachnoid space with the observation of cerebrospinal fluid outflow. The patient was placed in the supine position immediately after drug injection. Dermatomal level of sensorial block will be evaluated with pinprick test and modified Bormage scale was used to assess motor blockade. Surgery will be allowed after the achievement of sensorial block at the T10 level.

Monitoring and data collection Non-invasive blood pressure, heart rate (HR), peripheral oxygen saturation (SpO2) and continuous ECG monitorization will be obtained for all patients throughout the study via Mindray Bene View T8 (Shenzhen Mindray Bio-Medical Electronics Co., LTD, PR China. The QT interval will be measured automatically in lead II and calculation of the QTc interval was also achieved automatically with using Bazett's formula (QTc=QT/radqRR(sec)) from ECG monitorization. QT and QTc intervals will be measured and recorded in the following manner: before the anesthesia induction or subarachnoid injection (in group S), 1, 5, 10 minute after after endotracheal intubation or subarachnoid injection (in group S), and immediately after surgery. Presence of arrhythmia will also be recorded.

Patient characteristics including age, gender, height, weight, body mass index (BMI), comorbidity, ASA physical status classification and duration of surgery will be recorded. Moreover maximum sensory block level and motor block recovery time will be investigated in the group S. Also all cardiopulmonary adverse events will be evaluated including hypotension (decrease in mean blood pressure > 20%), bradycardia (HR < 50 beats/min) and hypoxemia (SpO2 < 90%).

Statistical analysis SPSS software package for Windows (Statistical Package for Social Sciences, version 22.0, SPSS Inc., Chicago, Illinois, USA) will be used for statistical analysis of study data. Quantitative variables were emitted as mean ± standard deviation (SD), whereas categorical variables as number of patients and percentage. Quantitative variables will be evaluated for distribution normality using the Kolmogorov-Smirnov/Shapiro-Wilk's test and independent student's t-test will be used to compare normally distributed variables between groups. To compare categorical variables chi-square or Fisher's exact test will be used. QT and QTc intervals within groups will be investigated with repeated measures analysis of variance and post hoc multiple comparisons will be performed by Bonferroni test. Sample size calculation was based on QTc interval. Based on a previous study, QTc interval was found 397.3±27.4 msec after spinal anesthesia in non-geriatric patients. Power analysis with α = 0.05 and β = 0.2 to detect an increase of at least 20 msec in QTc interval revealed that a min of 28 patients should be included in each group. A p value < 0.05 was considered to show a statistically significant result.

ELIGIBILITY:
Inclusion Criteria:

* patients who scheduled lower abdominal or extremity surgery and urological surgery older than 65 years were enrolled to the study.

Exclusion Criteria:

* any preoperative ECG abnormalities, QTc interval > 440 ms, family history of long QT syndome, use of any medications known to affect the QTc interval, serum electrolyte abnormalities, any contraindications for spinal anesthesia (e.g. coagulation disorders), unstable angina pektoris, chronic obstructive pulmonary disease, hepatic or renal failure, American Society of Anesthesiologists (ASA) physical classification status > III, pregnancy and obesity (BMI > 30).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — older than 65 years old
Enrollment: 58 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
QTc interval | before anesthesia induction or spinal anesthesia; 1, 5 and 10 minutes after endotrakeal intubation or spinal anesthesia; after extubation or surgery
  QTc interval on ECG calculated with Bazzets formula

SECONDARY OUTCOMES:
QT | before anesthesia induction or spinal anesthesia; 1, 5 and 10 minutes after endotrakeal intubation or spinal anesthesia; after extubation or surgery
  the time between the beginning of the QRS complex and the end of the T wave in electrocardiography

CONTACTS AND LOCATIONS:
Overall Officials: sinan uzman, Assoc. Prof., Study Director — Health Science University Haseki Training and Research Hospital
Locations (1):
- Health Science University, Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to drsinanuzman@yahoo.com

REFERENCES:
- [Background] Song JH, Yang C, Lee W, Kim H, Kim Y, Kim H. QTc interval prolongation due to spinal anesthesia in patients with and without diabetes: an observational study. BMC Anesthesiol. 2022 May 13;22(1):143. doi: 10.1186/s12871-022-01614-8. PMID 35562669